CLINICAL TRIAL: NCT00440739
Title: Etoricoxib With Flavoxate for Reducing Morphine Requirement After Transurethral Prostatectomy: A Factorial Randomized Controlled Trial
Brief Title: Etoricoxib With Flavoxate for Reducing Morphine Requirement After Transurethral Prostatectomy (TURP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Ethic committee Mahidol University, Mahidol University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SiEc 161/2548
Record Dates: First submitted 2006-02-02; First posted 2007-02-27 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2007-02

CONDITIONS: Pain
Keywords: postoperative pain, etoticoxib, etoricoxib; Pain relief after transurethral resection of prostate.
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Etoricoxib; Flavoxate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): 1=placebo
  Interventions: Drug: placebo
- 2 (Active Comparator): 2= etoricoxib
  Interventions: Drug: etoricoxib
- 3 (Active Comparator): 3=falvoxate
  Interventions: Drug: flavoxate
- 4 (Active Comparator): etoricoxib and flavoxate
  Interventions: Drug: etoricoxib, flavoxate

INTERVENTIONS:
Drug: etoricoxib — etoricoxib 120 mg
  Other Names: arcoxia
  Arms: 2
Drug: flavoxate — flavoxate 200 mg 3 times
  Other Names: urispas
  Arms: 3
Drug: etoricoxib, flavoxate — etoricoxib 120 mg once and flavoxate 200 mg 3 times
  Other Names: arcoxia; urispas
  Arms: 4
Drug: placebo — placebo once and placebo 3 times
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether etoricoxib, flavoxate, both are effective in the treatment postoperative pain after TURP.

The research hypothesis:

There is a difference in postoperative morphine consumption in the first 24 hours after transurethral prostatectomy between patients who received etoricoxib or flavoxate or both and placebo.

DETAILED DESCRIPTION:
Postoperative pain is still a significant problem for surgical patients. Conventional use of narcotics for postoperative pain relief is not without serious side effects such as respiratory depression and sedation.There are other alternatives for postoperative analgesia as NSAIDs especially COX2-inhibitors. For some specific operation such as TURP which Foley's catheter needed to be retained for a few days,urinary anti spasmodics may help the patients to be more comfortable.

Comparison(s): There is a difference in postoperative morphine consumption in the first 24 hours after transurethral prostatectomy between patients who received etoricoxib or flavoxate or both and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male patient ASA physical status I-III.
2. Scheduled for an elective TURP.
3. Body weight > or = 50 kg
4. Can operate a patient-controlled analgesia (PCA) device.

Exclusion Criteria:

1. History of asthma, acute rhinitis, nasal polyps, angioneurotic edema or urticaria following the administration of aspirin or other NSAIDs.
2. Known hypersensitivity to morphine.
3. History of hepatic dysfunction.
4. Creatinine clearance < 30ml/min.
5. History of bleeding tendency.
6. History of gastrointestinal bleeding or active peptic ulcer.
7. Known case of inflammatory bowel disease.
8. Patient with severe heart failure.
9. History of coronary artery disease or cerebrovascular disease.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2005-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The patients' total amount of morphine requirement in the first 24 hour. | 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok 10700, Thailand
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand